CLINICAL TRIAL: NCT02846688
Title: Gene Expression Profiling in Human Gastric Intestinal Metaplasia Mucosa and Duodenal Mucosa.
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Gene Expression Profiling in Human Gastric Intestinal Metaplasia Mucosa and Duodenal Mucosa, Shandong University
Other Study IDs: 2015SDU-QILU-G05
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Gene Expression Profiling; Gastric Intestinal Metaplasia; Duodenum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The metagenome was obtained from biopsy specimen.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To analyze the genome pattern in human gastric Intestinal Metaplasia Mucosa and duodenal Mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for gastroendoscopy examination

Exclusion Criteria:

* Esophageal, gastric or duodenal cancer or other malignancy History of upper GI tract surgery Coagulopathy or bleeding disorders Allergy to fluorescein sodium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective patients scheduled for pCLE examination at Qilu Hospital, Shandong University
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Gene Expression Profiling in Human Gastric Intestinal Metaplasia Mucosa and Duodenal Mucosa | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: li yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China